CLINICAL TRIAL: NCT00212953
Title: Ontario Prehospital Advanced Life Support (OPALS) Study Phase III Cardiac Arrest and Critical Care Sub-Studies - Chest Pain Sub-Study, Respiratory Sub-Study, and Major Trauma Sub-Study
Brief Title: OPALS Critical Care Sub-Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Ian Stiell, Principal Investigator, Ottawa Hospital Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1997576-01H
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac Arrest
Keywords: Chest Pain,; Shortness of breath,; Injury,; Trauma
MeSH Terms: conditions — Heart Arrest; Chest Pain; Dyspnea; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Advanced Life Support

SUMMARY:
The purpose of the study is to evaluate the incremental benefit of a full advanced life support EMS program on the outcomes of chest pain, respiratory and major trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Chest Pain Sub-Study: Adult patients with a complaint of chest pain of an acute nature transported to hospital by ambulance. Patients with a complaint of pain in arms, neck or jaw if consistent with myocardial ischemia. Patients must have an ambulance return code of prompt, urgent, or no patient carried.
* Respiratory Sub-Study: Adult patients with a chief complaint of shortness of breath defined as ACR codes of Respiratory Failure, Shortness of Breath NYD, Pulmonary Edema (CHF), Asthma and had either prehospital assisted ventilation or abnormal respiratory rates (>=24 or <=10)
* Major Trauma Sub-Study: Adult patients who have suffered an injury from any mechanism with an Injury Severity Score of >12 who have been transported to hospital by land ambulance, and who have been entered into the Ontario Trauma Registry (OTR) Comprehensive Data Set.

Exclusion Criteria:

* All Sub-Studies:
* Patients under the age of 16
* Patients who are vital signs absent prior to EMS arrival.
* Chest Pain Sub-Study:
* Patients suffering primarily from respiratory distress, respiratory failure, pulmonary edema, asthma, palpitations or epigastric pain. pain

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21000
Dates: Start 1997-03; Study Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Survival to discharge

SECONDARY OUTCOMES:
Generic Quality of Life
Disease Specific Quality of Life CPC Score and FIM Score
Performance of ALS Procedures
Response Time Intervals
Length of Stay in Hospital
Length of Stay in Critical Care Units
Ventilator time
Disease Specific Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — OHRI
Locations (11):
- Canada (11):
  - Cambridge Base Hospital, Cambridge, Ontario
  - Sudbury Base Hospital, Greater Sudbury, Ontario
  - Kingston Base Hospital, Kingston, Ontario
  - London Base Hospital, London, Ontario
  - Halton Base Hospital, Mississauga, Ontario
  - Niagara Falls Base Hospital, Niagara Falls, Ontario
  - Ottawa Base Hospital, Ottawa, Ontario
  - Peterborough Base Hospital, Peterborough, Ontario
  - Lambton Base Hospital, Sarnia, Ontario
  - Thunder Bay Base Hospital, Thunder Bay, Ontario
  - Windsor Base Hospital, Windsor, Ontario